CLINICAL TRIAL: NCT00002651
Title: Intermittent Androgen Deprivation in Patients With Stage D2 Prostate Cancer, Phase III
Brief Title: SWOG-9346, Hormone Therapy in Treating Men With Stage IV Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NCIC Clinical Trials Group (Network); Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network); European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000064184; SWOG-9346; CAN-NCIC-PR8; CALGB-9594; ECOG-S9346; EORTC-30985; CAN-NCIC-JPR8; INT-0162
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Goserelin; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Consolidation arm I (Active Comparator): Patients continue CAD therapy comprising goserelin subcutaneously once a month and oral bicalutamide once daily. Treatment continues in the absence of disease progression.
  Interventions: Drug: bicalutamide; Drug: goserelin acetate
- Consolidation arm II (Experimental): Patients undergo observation in the absence of rising prostate-specific antigen (PSA) or clinical symptoms of progressive disease. Patients with rising PSA or progressive disease begin CAD therapy as in consolidation arm I. Patients whose PSA normalizes after 8 courses return to observation. Patients whose PSA does not normalize after 8 courses continue CAD therapy.
  Interventions: Drug: bicalutamide; Drug: goserelin acetate; Other: clinical observation

INTERVENTIONS:
Drug: bicalutamide — Given orally
Drug: goserelin acetate — Given subcutaneously
Other: clinical observation — Patients undergo observation in the absence of rising prostate-specific antigen (PSA) or clinical symptoms of progressive disease.
  Arms: Consolidation arm II

SUMMARY:
RATIONALE: Testosterone can stimulate the growth of prostate cancer cells. Hormone therapy may be effective treatment for prostate cancer. It is not yet known which regimen of hormone therapy is most effective for stage IV prostate cancer.

PURPOSE: This randomized phase III trial is studying two different regimens of hormone therapy and comparing how well they work in treating men with stage IV prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the survival of patients with metastatic stage IV prostate cancer responsive to combined androgen-deprivation therapy (CAD) treated with intermittent vs continuous CAD.
* Compare the effects of these treatment regimens on impotence, libido, and vitality/fatigue as well as the physical and emotional well-being of these patients.

Secondary

* Compare general symptoms, role functioning, global perception of quality of life, and social functioning of patients treated with these regimens.
* Assess prostate-specific antigen (PSA) levels after continuous CAD administered before randomization and evaluate PSA changes throughout randomized treatment of these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to SWOG performance status (0-1 vs 2), severity of disease (minimal vs extensive), and prior hormonal therapy (neoadjuvant hormonal therapy vs finasteride vs neither).

* Induction therapy: Patients receive combined androgen-deprivation (CAD) therapy comprising goserelin subcutaneously once a month and oral bicalutamide once daily for 8 courses (7 months).
* Consolidation therapy: Patients are randomized to 1 of 2 consolidation regimens.

  * Arm I (continuous CAD therapy): Patients continue CAD therapy as in induction therapy. Treatment continues in the absence of disease progression.
  * Arm II (intermittent CAD therapy): Patients undergo observation in the absence of rising prostate-specific antigen (PSA) or clinical symptoms of progressive disease. Patients with rising PSA or progressive disease begin CAD therapy as in induction therapy. Patients whose PSA normalizes after 8 courses return to observation. Patients whose PSA does not normalize after 8 courses continue CAD therapy.

Quality of life is assessed before induction therapy, at 3 months (before consolidation therapy), and then at 9 and 15 months.

Patients are followed every 6-12 months for at least 10 years.

PROJECTED ACCRUAL: Approximately 1,500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the prostate

  * Metastatic stage IV (stage D2)

    * Any number of bone metastases by bone scan allowed
    * Unequivocal visceral organ metastases (liver, brain, or lung) allowed
  * No suspected second primary tumors unless metastases are histologically confirmed, including special stains (e.g., prostate specific antigen [PSA] and prostatic alkaline phosphatase [PAP])
* For entry into late induction therapy:

  * No more than 1 month from the beginning of antiandrogen therapy to the beginning of luteinizing hormone-releasing hormone (LHRH) agonist therapy
  * No more than 6 months since initiation of current combined androgen-deprivation therapy (LHRH agonist and antiandrogen)
  * The effectiveness of the current depot LHRH agonist would not extend beyond 8 months after initiation of combined androgen therapy
* PSA at least 5 ng/mL
* No acute spinal cord compression

PATIENT CHARACTERISTICS:

Age:

* Adult

Performance status:

* SWOG 0-2

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Recovered from any major infection
* No active medical illness that would preclude study or limit survival
* No other malignancy within the past 5 years except:

  * Adequately treated basal cell or squamous cell skin cancer
  * Adequately treated carcinoma in situ of the bladder
  * Adequately treated other superficial cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biological response modifier therapy

Chemotherapy:

* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* More than 1 year since any prior neoadjuvant or adjuvant hormonal therapy for a duration of no more than 4 months

  * Single or combination therapy allowed
* More than 1 year since prior finasteride for prostate cancer for a duration of no more than 9 months (less than 6 months for benign prostatic hypertrophy)
* Prior or concurrent megestrol for hot flashes allowed
* No other concurrent hormonal therapy

Radiotherapy:

* No concurrent radiotherapy other than palliation of painful bone metastases

Surgery:

* No prior bilateral orchiectomy
* Recovered from any prior major surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3040 (Actual)
Dates: Start 1995-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hadi A. Hussain, MD, Study Chair — University of Michigan Rogel Cancer Center; Bryan J. Donnelly, MD, FRCSC, MSC, Study Chair — Tom Baker Cancer Centre - Calgary; Eric J. Small, MD, Study Chair — University of California, San Francisco; George Wilding, MD, Study Chair — University of Wisconsin, Madison; Atif Akdas, MD, Study Chair — Marmara University Hospital
Locations (14):
- Canada (14):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - CHUS-Hopital Fleurimont, Sherbrooke, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Tangen CM, Hussain MH, Higano CS, Eisenberger MA, Small EJ, Wilding G, Donnelly BJ, Schelhammer PF, Crawford ED, Vogelzang NJ, Powell IJ, Thompson IM Jr. Improved overall survival trends of men with newly diagnosed M1 prostate cancer: a SWOG phase III trial experience (S8494, S8894 and S9346). J Urol. 2012 Oct;188(4):1164-9. doi: 10.1016/j.juro.2012.06.046. Epub 2012 Aug 22. PMID 22921015
- [Background] Hussain M, Tangen CM, Higano CS, et al.: Improved overall survival (OS) of patients (pts) with new metastatic prostate cancer (pca): better efficacy or stage migration? Data from SWOG: S9346 and 8894. [Abstract] 2010 Genitourinary Cancers Symposium, March 5-7, 2010, San Francisco, California. A-30, 2010.
- [Background] Hussain M, Goldman B, Tangen C, Higano CS, Petrylak DP, Wilding G, Akdas AM, Small EJ, Donnelly BJ, Sundram SK, Burch PA, Dipaola RS, Crawford ED. Prostate-specific antigen progression predicts overall survival in patients with metastatic prostate cancer: data from Southwest Oncology Group Trials 9346 (Intergroup Study 0162) and 9916. J Clin Oncol. 2009 May 20;27(15):2450-6. doi: 10.1200/JCO.2008.19.9810. Epub 2009 Apr 20. PMID 19380444
- [Background] Goldman B, Hussain M, Tangen C, et al.: Prostate-specific antigen progression (PSA-P) as a predictor of overall survival (OS) in patients (pts) with metastatic prostate cancer (PC): data from S9346 and S9916. [Abstract] American Society of Clinical Oncology 2008 Genitourinary Cancers Symposium, Feb 14-16, 2008, San Francisco, CA. A-165, 2008.
- [Background] Hussain MH, Goldman B, Tangen CM, et al.: Use of prostate-specific antigen progression (PSA-P) to predict overall survival (OS) in patients (pts) with metastatic prostate cancer (PC): data from S9346 and S9916. [Abstract] J Clin Oncol 26 (Suppl 15): A-5015, 2008.
- [Result] Hussain M, Tangen CM, Higano CS, et al.: Intermittent (IAD) versus continuous androgen deprivation (CAD) in hormone sensitive metastatic prostate cancer (HSM1PC) patients (pts): results of S9346 (INT-0162), an international phase III trial. [Abstract] J Clin Oncol 30 (Suppl 15): A-4, 2012.
- [Result] Moinpour C, Berry DL, Ely B, et al.: Preliminary quality-of-life outcomes for SWOG-9346: Intermittent androgen deprivation in patients with hormone-sensitive metastatic prostate cancer (HSM1PC)-phase III. [Abstract] J Clin Oncol 30 (Suppl 15): A-4571, 2012.
- [Result] Hussain M, Tangen CM, Higano C, Schelhammer PF, Faulkner J, Crawford ED, Wilding G, Akdas A, Small EJ, Donnelly B, MacVicar G, Raghavan D; Southwest Oncology Group Trial 9346 (INT-0162). Absolute prostate-specific antigen value after androgen deprivation is a strong independent predictor of survival in new metastatic prostate cancer: data from Southwest Oncology Group Trial 9346 (INT-0162). J Clin Oncol. 2006 Aug 20;24(24):3984-90. doi: 10.1200/JCO.2006.06.4246. PMID 16921051
- [Result] Tangen CM, Hussain M, Wilding G, et al.: Determinants of prostate specific antigen (PSA) normalization in prostate cancer (PCa) patients (pts) treated with androgen deprivation (AD) on Southwest Oncology Group (SWOG) study 9346 (INT-0162). [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1591, 2003.
- [Derived] Hershman DL, Unger JM, Wright JD, Ramsey S, Till C, Tangen CM, Barlow WE, Blanke C, Thompson IM, Hussain M. Adverse Health Events Following Intermittent and Continuous Androgen Deprivation in Patients With Metastatic Prostate Cancer. JAMA Oncol. 2016 Apr;2(4):453-61. doi: 10.1001/jamaoncol.2015.4655. PMID 26720308
- [Derived] Eggener S. Commentary on "Intermittent versus continuous androgen deprivation in prostate cancer." Hussain M, Tangen CM, Berry DL, Higano CS, Crawford ED, Liu G, Wilding G, Prescott S, Kanaga Sundaram S, Small EJ, Dawson NA, Donnelly BJ, Venner PM, Vaishampayan UN, Schellhammer PF, Quinn DI, Raghavan D, Ely B, Moinpour CM, Vogelzang NJ, Thompson IM Jr, University of Michigan, Division of Hematology/Oncology, Ann Arbor, MI. N Engl J Med 2013; 368(14):1314-25. doi: 10.1056/NEJMoa1212299. Urol Oncol. 2014 Aug;32(6):936-7. doi: 10.1016/j.urolonc.2014.01.009. PMID 25087673
- [Derived] Hussain M, Tangen CM, Berry DL, Higano CS, Crawford ED, Liu G, Wilding G, Prescott S, Kanaga Sundaram S, Small EJ, Dawson NA, Donnelly BJ, Venner PM, Vaishampayan UN, Schellhammer PF, Quinn DI, Raghavan D, Ely B, Moinpour CM, Vogelzang NJ, Thompson IM Jr. Intermittent versus continuous androgen deprivation in prostate cancer. N Engl J Med. 2013 Apr 4;368(14):1314-25. doi: 10.1056/NEJMoa1212299. PMID 23550669

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Androgen Deprivation (CAD): Patients receive goserelin 3.6 mg subcutaneously once a month and oral bicalutamide 50 mg once daily for 7 months.
- Continuous Hormonal Therapy: Patients continue to receive goserelin 3.6 mg subcutaneously once a month and oral bicalutamide 50 mg once daily until progression of disease
- Intermittent Hormonal Therapy: Patients are cycled between observation periods and Combined Androgen Deprivation (CAD) periods based on PSA results. Patients undergo observation in the absence of rising prostate-specific antigen (PSA) or clinical symptoms of progressive disease. Patients with rising PSA or progressive disease begin CAD therapy (goserelin 3.6 mg subcutaneously once a month and oral bicalutamide 50 mg once daily ). Patients whose PSA normalizes after 8 cycles of CAD treatment return to observation. Patients whose PSA does not normalize after 8 cycles of CAD treatment continue CAD therapy until progression (1 cycle of CAD treatment = 7 months with 8 injections. There are 2 injections in the first month on Days 1 and 29).
Period: Induction
Arm/Group | Combined Androgen Deprivation (CAD) | Continuous Hormonal Therapy | Intermittent Hormonal Therapy
Started | 3040 | 0 | 0
Eligible | 2950 | 0 | 0
Eligible and Began Protocol Therapy | 2950 | 0 | 0
Completed | 1697 | 0 | 0
Not Completed | 1343 | 0 | 0
Not completed — Adverse Event | 44 | 0 | 0
Not completed — Refusal unrelated to adverse event | 50 | 0 | 0
Not completed — Progression/relapse | 274 | 0 | 0
Not completed — Death | 62 | 0 | 0
Not completed — Other | 823 | 0 | 0
Not completed — not eligible | 90 | 0 | 0
Period: Consolidation and Randomization
Arm/Group | Combined Androgen Deprivation (CAD) | Continuous Hormonal Therapy | Intermittent Hormonal Therapy
Started | 0 | 867 (After induction,patients with stable or declining PSA (≤ 4.0 ng/mL) were eligible for randomization) | 882 (After induction,patients with stable or declining PSA (≤ 4.0 ng/mL) were eligible for randomization)
Eligible | 0 | 765 | 770
Assessable for Toxicity (Patients with no AE evaluations, received wrong protocol arm, or received non-protocol trt excluded) | 0 | 732 | 702
Completed | 0 | 29 | 22
Not Completed | 0 | 838 | 860
Not completed — Adverse Event | 0 | 36 | 14
Not completed — Refusal unrelated to adverse event | 0 | 53 | 75
Not completed — Progression/relapse | 0 | 295 | 298
Not completed — Death | 0 | 38 | 48
Not completed — Other | 0 | 314 | 313
Not completed — not eligible | 0 | 102 | 112

BASELINE CHARACTERISTICS:
Population: Randomized and eligible patients (After induction, Patients with stable or declining PSA levels of 4.0 ng per milliliter or lower at months 6 and 7 were eligible for randomization).
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Hormonal Therapy | Intermittent Hormonal Therapy | Total
Number analyzed (Participants) | 765 | 770 | 1535
Age, Continuous [Median (Full Range); unit: years] | 70 [39 to 92] | 70 [39 to 97] | 70 [39 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 765 | 770 | 1535
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 23 | 40
  Not Hispanic or Latino | 571 | 564 | 1135
  Unknown or Not Reported | 177 | 183 | 360
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 5 | 8 | 13
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 93 | 94 | 187
  White | 507 | 519 | 1026
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 154 | 144 | 298

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Non-inferiority test to determine if intermittent combined androgen deprivation (CAD) overall survival is not substantially worse than continuous CAD overall survival. Specifically, the trial is designed for a one-sided test of the hypothesis that the hazard ratio of intermittent CAD to continuous CAD is 1.2. The assumptions used to compute the trial size are an overall type I error rate of 0.05 and a type II error of 0.10 (power = 0.9).
Time Frame: Up to 15 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Consolidation Arm I | Consolidation Arm II
Number analyzed (Participants) | 765 | 770
years | 5.8 [5.3 to 6.4] | 5.1 [4.8 to 5.5]
Statistical Analysis 1: Comparison: Consolidation Arm I vs Consolidation Arm II; Test type: Non-Inferiority or Equivalence — The overall type I error rate used is 0.05. The type II error rate is 0.10 (power = 0.9). The trial planned for a one-sided test of the hypothesis that the hazard ratio of intermittent CAD to continuous CAD is 1.2. A hazard ratio of 1.0 was used as the specific alternative in the trial size computations. Thus, rejection of the hypothesis will be evidence against the possibility that the intermittent CAD hazard ratio is larger than the continuous CAD hazard ratio by 20% or more; p = 0.15, Regression, Cox; Hazard Ratio (HR) = 1.10, 90% CI 2-sided [0.99 to 1.23]

2. Primary Outcome: Physical Functioning as Measured by the SF-36
Description: This outcome was scored on a scale of 0 to 100, with higher scores indicating better functioning. Change from Baseline in SF-36 Score at 3 Months
Time Frame: 3 months
Population: Only eligible patients with a usable form set for Physical Functioning portion of the SF-36 both at baseline and 3 months were included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Hormonal Therapy | Intermittent Hormonal Therapy
Number analyzed (Participants) | 469 | 475
units on a scale | -1.74 (0.7366) | 0.09 (0.8084)
Statistical Analysis 1: Comparison: Continuous Hormonal Therapy vs Intermittent Hormonal Therapy; Test type: Superiority or Other; p = 0.09, t-test, 2 sided — The type I error rate used was 0.005 in an attempt to adjust for multiple primary scores being tested.The type II error rate used was 0.10 (power = 0.9); Mean Difference (Net) = 1.83, 95% CI 2-sided [-0.31 to 3.97]

3. Primary Outcome: Emotional Functioning as Measured by the SF-36 Mental Health Inventory
Description: as for outcome 2
Time Frame: 3 months
Population: Only eligible patients with a usable form set for SF-36 Mental Health Inventory both at baseline and 3 months were included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Hormonal Therapy | Intermittent Hormonal Therapy
Number analyzed (Participants) | 471 | 479
units on a scale | -0.95 (0.6804) | 1.92 (0.7241)
Statistical Analysis 1: Comparison: Continuous Hormonal Therapy vs Intermittent Hormonal Therapy; Test type: Superiority or Other; p = 0.003, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 2.88, 95% CI 2-sided [1.00 to 4.76]

4. Primary Outcome: Erectile Dysfunction
Description: This outcome was assessed by having patients report whether they had erectile dysfunction (a score of 1) or no erectile dysfunction (a score of 0). This analysis looks at change from Baseline to 3 Months.
Time Frame: 3 months
Population: Only eligible patients with a usable answers regarding erectile dysfunction both at baseline and 3 months were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Continuous Hormonal Therapy | Intermittent Hormonal Therapy
Number analyzed (Participants) | 450 | 466
percentage of participants | 2 | -7
Statistical Analysis 1: Comparison: Continuous Hormonal Therapy vs Intermittent Hormonal Therapy; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -10, 95% CI 2-sided [-14 to -5]

5. Primary Outcome: High Libido
Description: This outcome was assessed by having patients report whether their interest in sexual activities was very high, high, or moderate (a score of 1) or low or very low (a score of 0). This outcome measure is reporting a change from baseline in the percentage of participants with High Libido at 3 months. "High Libido" is defined as very high, high or moderate interest in sexual activities.
Time Frame: 3 months
Population: Only eligible patients with a usable answers regarding libido both at baseline and 3 months were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Continuous Hormonal Therapy | Intermittent Hormonal Therapy
Number analyzed (Participants) | 45 | 68
percentage of participants | -2 | 16
Statistical Analysis 1: Comparison: Continuous Hormonal Therapy vs Intermittent Hormonal Therapy; Test type: Superiority or Other; p = 0.04, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 18, 95% CI 2-sided [1 to 36]

6. Primary Outcome: Vitality
Description: This outcome was scored on a scale of 0 to 100, with higher scores indicating better functioning. This analysis looks at mean change from Baseline score to 3 Months.
Time Frame: 3 months
Population: Only eligible patients with a usable form set for Vitality both at baseline and 3 months were included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Hormonal Therapy | Intermittent Hormonal Therapy
Number analyzed (Participants) | 446 | 465
units on a scale | -1.42 (0.7379) | -0.11 (0.8154)
Statistical Analysis 1: Comparison: Continuous Hormonal Therapy vs Intermittent Hormonal Therapy; Test type: Superiority or Other; p = 0.23, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 1.32, 95% CI 2-sided [-0.83 to 3.46]

7. Other Pre Specified Outcome: Global Perception of Quality of Life
Time Frame: 15 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Social Functioning
Description: Mean of the change in social functioning from randomization
Time Frame: 15 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Role Functioning
Description: Mean of the change in role functioning from randomization
Time Frame: 15 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: General Symptoms
Time Frame: 15 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 10 years after registration to Induction
Description: Participants were monitored for toxicity every 3 months while on protocol therapy or at more frequent intervals appropriate for that participant, as judged by the treating physician.
Arm/Group | Continuous Hormonal Therapy | Intermittent Hormonal Therapy
Serious Adverse Events (participants affected / at risk) | 19/732 | 10/702
Other Adverse Events (participants affected / at risk) | 665/732 | 609/702
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Hormonal Therapy (N=732) | Intermittent Hormonal Therapy (N=702)
Cardiac ischemia/infarction (Cardiac disorders) | 6 | 2
Cardiovascular-other (Cardiac disorders) | 2 | 1
LVEF decrease/CHF (Cardiac disorders) | 1 | 1
Flu-like symptoms-other (General disorders) | 5 | 3
Second primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular ischemia (Nervous system disorders) | 1 | 1
Lung-other (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusions (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemorrhage-other (Vascular disorders) | 1 | 0
Thrombosis/embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Hormonal Therapy (N=732) | Intermittent Hormonal Therapy (N=702)
Anemia (Blood and lymphatic system disorders) | 86 | 85
Constipation/bowel obstruction (Gastrointestinal disorders) | 81 | 55
Diarrhea without colostomy (Gastrointestinal disorders) | 93 | 79
Nausea (Gastrointestinal disorders) | 54 | 38
Fatigue/malaise/lethargy (General disorders) | 381 | 364
Pain-other (General disorders) | 140 | 131
Alkaline phosphatase increase (Investigations) | 58 | 95
Creatinine increase (Investigations) | 107 | 87
SGOT (AST) increase (Investigations) | 49 | 70
Weight gain (Investigations) | 60 | 33
Hyperglycemia (Metabolism and nutrition disorders) | 85 | 91
Arthralgia (Musculoskeletal and connective tissue disorders) | 92 | 63
Bone pain (Musculoskeletal and connective tissue disorders) | 239 | 272
Myalgia (Musculoskeletal and connective tissue disorders) | 44 | 42
Dizziness/light headedness (Nervous system disorders) | 44 | 38
Sensory neuropathy (Nervous system disorders) | 111 | 95
Weakness (motor neuropathy) (Nervous system disorders) | 75 | 61
Anxiety/agitation (Psychiatric disorders) | 41 | 41
Depression (Psychiatric disorders) | 107 | 96
Insomnia (Psychiatric disorders) | 141 | 123
Libido loss (Psychiatric disorders) | 262 | 226
Urinary frequency/urgency (Renal and urinary disorders) | 141 | 147
Erectile impotence (Reproductive system and breast disorders) | 304 | 256
Gynecomastia (Reproductive system and breast disorders) | 181 | 158
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 43
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 109 | 116
Rash/desquamation (Skin and subcutaneous tissue disorders) | 81 | 65
Sweating (Skin and subcutaneous tissue disorders) | 245 | 176
Hot flashes (Vascular disorders) | 511 | 440
Hypertension (Vascular disorders) | 37 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No